CLINICAL TRIAL: NCT00524550
Title: Effect of Moderate Alcohol Consumption on Postprandial Insulin Secretion, Appetite Regulation, Glucose Homeostasis and Insulin Resistance.
Brief Title: Postprandial Insulin Secretion and Appetite Regulation After Moderate Alcohol Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Responsible Party: henk FJ Hendriks, TNO Quality of life
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: P7573; Alcohol Research 21
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: Moderate alcohol consumption; insulin secretion; insulin sensitivity; Beta-cell function; Adiponectin; Appetite; Satiety; Alcohol-induced gene expression; Endocannabinoids; Glucose metabolism; Lipid metabolism; Ratio HMW/total adiponectin; Appetite regulation; Alcohol-induced adiponectin increase
MeSH Terms: conditions — Insulin Resistance | interventions — Ethanol; Economics

INTERVENTIONS:
Dietary Supplement: moderate alcohol consumption — drinking commercially available alcohol-free beer or beer (26 grams of alcohol per day), for three weeks

SUMMARY:
A body of epidemiologic studies show that moderate alcohol consumption is associated with a protective effect against type 2 diabetes. The importance of both insulin sensitivity and insulin secretion in the pathogenesis of glucose intolerance and diabetes type 2 is widely recognized. Clinical studies show improved insulin sensitivity after a period of alcohol consumption compared to abstention. However, postprandial insulin secretion and beta-cell function after a period of moderate alcohol consumption have scarcely been addressed in published literature.

When consumed as an aperitif or with a meal, alcohol is generally expected to stimulate appetite and food intake and thus might be a risk factor for over consumption and obesity. However the physiological mechanisms for this observed effect are not well understood. Furthermore, previous studies lacked a link between physiological parameters and subjective parameters of satiety.

DETAILED DESCRIPTION:
Objective:

Primary objectives are to study the effects of moderate alcohol consumption on

* Postprandial insulin secretion and pancreatic beta-cell function
* Physiological and subjective parameters related to satiety and appetite

Secondary objectives are to study the effects of moderate alcohol consumption on

* Miscellaneous markers of glucose homeostasis and insulin sensitivity
* Kinetics of alcohol-induced increase of adiponectin

A tertiary objective is to study the effects of moderate alcohol consumption on

* Gene expression in subcutaneous adipose tissue in normal-weight pre menopausal women with normal fasting plasma glucose.

Study design: Randomized, partially controlled, open label, cross-over study with a one week wash-out preceding each treatment period

Study population: 24 apparently healthy pre menopausal Caucasian women with fasting blood glucose <6.1 mmol/L, aged 20 - 44 years at inclusion of the study, with a BMI of 19 - 25 kg/m2, who use oral contraceptives will participate in the study.

Intervention: Participants will drink daily a test substance for three weeks (2 cans of Amstel beer per day; 66 cL ~ 26 gram alcohol) followed by a reference substance (2 cans of Amstel alcohol-free beer per day; 66 cL < 0.5 gram of alcohol) for three weeks or vice versa. Both treatments are preceded by a one-week wash-out period in which no alcohol is consumed.

ELIGIBILITY:
Inclusion Criteria:

* Apparently Females between 20 - 44 years of age
* Using oral contraceptives for >3 months (only phase 1 or 2 oral contraceptives)
* Normal fasting glucose levels as indicated by venous fasting plasma glucose levels < 6.1 mmol/L
* Alcohol consumption more or equal then 5 and less than 22 glasses/week
* Body Mass Index (BMI) between 19 and 25 kg/m2

Exclusion Criteria:

* Having the intention to become pregnant, to be pregnant or to lactate during the study
* Having a history of medical or surgical events that may significantly affect the study outcome including metabolic or endocrine disease, gastro-intestinal disorder, or eating behavior disorders such as anorexia/bulimia disorders
* Having a family history of alcoholism
* Smoking
* Reported use of any soft or hard drugs
* Reported unexplained weight loss or gain of > 3 kg in the month prior to the screening

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Pancreatic beta-cell function | 3 weeks of treatment preceded by a 1-week wash-out
Satiety | 3 weeks of treatment preceded by a 1-week wash-out

SECONDARY OUTCOMES:
Kinetics of adiponectin | 3 weeks of treatment preceded by a 1-week wash-out

CONTACTS AND LOCATIONS:
Overall Officials: Henk FJ Hendriks, PhD, Principal Investigator — Hendriks HFJ
Locations (1):
- TNO Quality of Life, Zeist, Utrecht, Netherlands

REFERENCES:
- [Result] Joosten MM, Balvers MG, Verhoeckx KC, Hendriks HF, Witkamp RF. Plasma anandamide and other N-acylethanolamines are correlated with their corresponding free fatty acid levels under both fasting and non-fasting conditions in women. Nutr Metab (Lond). 2010 Jun 14;7:49. doi: 10.1186/1743-7075-7-49. PMID 20546561
- [Derived] Joosten MM, Schrieks IC, Hendriks HF. Effect of moderate alcohol consumption on fetuin-A levels in men and women: post-hoc analyses of three open-label randomized crossover trials. Diabetol Metab Syndr. 2014 Feb 18;6(1):24. doi: 10.1186/1758-5996-6-24. PMID 24548643
- [Derived] Joosten MM, Witkamp RF, Hendriks HF. Alterations in total and high-molecular-weight adiponectin after 3 weeks of moderate alcohol consumption in premenopausal women. Metabolism. 2011 Aug;60(8):1058-63. doi: 10.1016/j.metabol.2011.01.001. Epub 2011 Feb 24. PMID 21353262
- See also: publication — http://www.nutritionandmetabolism.com/content/7/1/49